CLINICAL TRIAL: NCT05233007
Title: Molecular Characterisation of Serial Tumour Samples and Their Correlation With Circulating Biomarkers and Other Biospecimens Taken During the Clinical Course of Patients Receiving Treatment for Upper Gastrointestinal Carcinomas.
Brief Title: Upper GI Serial Tumour Biopsies
Status: Suspended | Type: Observational
Why Stopped: To explore alternative funding streams
Sponsor: The Christie NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CFTSp209; 21/WM/0264 (Other: West Midlands - South Birmingham REC); 304901 (Other: IRAS)
Record Dates: First submitted 2022-01-31; First posted 2022-02-10 (Actual); Last update posted 2024-02-08 (Actual); Status verified 2024-02

CONDITIONS: Oesophageal Cancer; Gastric Cancer
MeSH Terms: conditions — Esophageal Neoplasms; Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Tumour biopsies, whole blood and blood products
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All participants: All eligible, consented participants, will be asked to give blood, tissue, and other biospecimens for research purposes
  Interventions: Procedure: Minor endoscopic biopsy

INTERVENTIONS:
Procedure: Minor endoscopic biopsy — As per standard of care

SUMMARY:
This is a prospective translational research study in which tumour samples, blood samples and other biospecimens will be requested from patients with locally advanced or metastatic malignant oesophageal and gastric carcinoma. There are two parts to the study:

* Part A - evaluation of serial tumour biopsies
* Part B - evaluation of circulating biomarkers and other biospecimens

DETAILED DESCRIPTION:
This is a prospective, non-randomised, non-interventional, translational research study in which patients with locally advanced or metastatic oesophageal and gastric carcinoma will be asked to donate tissue, blood and other available biospecimens for translational and biomarker research. This is an exploratory biomarker study to generate preliminary data for future research projects incorporating identified aberrations.

The overall aims of the study are to employ serial tumour biopsies, blood borne biomarkers and other biospecimens to investigate mechanisms of resistance to systemic therapy and develop predictive biomarkers of this resistance in patients with locally advanced and metastatic malignant oesophageal and gastric carcinoma. Blood biomarkers will include enumeration and characterisation of circulating blood cell subtypes, as well as the evaluation of circulating cell-free proteins and nucleic acids. Other biospecimens include urine, stool and hair follicle samples that the patient is willing to donate for research purposes, and ascitic, pleural, pericardial or cerebral spinal fluid, available to collect as part of clinically indicated procedures (standard care) and surplus to routine clinical requirements. These other biospecimens would be stored at the Biobank.

ELIGIBILITY:
Inclusion Criteria:

1. Age of 18 years or more.
2. Patients must have given written informed consent.
3. Evidence of locally advanced or metastatic oesophageal and gastric carcinoma, i.e. stage III or IV disease.
4. Accessible tumour that can be safely biopsied using radiological or surgical techniques (if consenting to part A).
5. Full blood count and coagulation tests within acceptable parameters (if consenting to part A).

Exclusion Criteria:

1. Inability to provide informed consent.
2. History of significant bleeding disorder (patients on anticoagulation are eligible if the anticoagulation can be safely managed to allow fresh tumour biopsies and blood sampling).
3. History of HIV, Hepatitis B/C or other transmissible human disease.
4. Any conditions where research biopsies or blood sampling may increase risk of complications for the patient and/or investigator, including high risk groups such as intravenous drug users.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Upper GI cancer patients, as determined by practicing oncologist
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2022-01-25 (Actual); Primary Completion 2028-10 (Estimated); Study Completion 2028-10 (Estimated)

PRIMARY OUTCOMES:
Determine levels of circulating biomarkers in upper GI cancer patients | 20 years
  To determine detectable levels of circulating biomarkers in patients with locally advanced and metastatic oesophageal and gastric carcinoma.
Correlating levels of biomarkers | 20 years
  To correlate circulating biomarker characteristics with serial tumour biopsies.
Predicting treatment resistance to anti-cancer therapy | 20 years
  To correlate sequencing/profiling data with clinical outcome data, including prognosis and response to systemic therapy.

CONTACTS AND LOCATIONS:
Locations (1):
- The Christie Hospital NHS Foundation Trust, Manchester, Greater Manchester, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided